CLINICAL TRIAL: NCT06298370
Title: The Efficacy of Combined Intrathecal Morphine and Pericapsular Nerve Group (PENG) Block on Postoperative Pain and Recovery Quality in Anterior Hip Arthroplasty: A Prospective, Double-blind, Randomized Clinical Trial
Brief Title: The Efficacy of Combined Intrathecal Morphine and PENG Block on Postoperative Pain in Hip Arthroplasty
Acronym: PENG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Saadet Oztop, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PENG study
Record Dates: First submitted 2024-02-03; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain Management
Keywords: Postoperative pain; Intrathecal morphine; Intrathecal bupivacaine; Hip arthroplasty; Pericapsular nerve group block
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Morphine

STUDY DESIGN:
Intervention Model Description: prospective, double-blind, randomized clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group P (Active Comparator): Patients in this group will undergo ultrasound-guided block using a linear or convex ultrasound probe in the supine position before intrathecal bupivacaine. The block procedure will involve the use of a local anesthetic solution (10-20 ml of 0.25% bupivacaine and 2 mg dexamethasone) and a 22 Gauche 80 mm block needle. Subsequently, intrathecal drug will be administered at the L3-L4 intervertebral level with 10-15 mg of bupivacaine while the patient is in a sitting position.
  Interventions: Drug: Pericapsular nerve group block plus intrathecal bupivacaine
- Group M (Active Comparator): Patients will receive intrathecal bupivacaine plus morphine without Pericapsular Nerve Group block. Intrathecal drugs will be administered at the L3-L4 intervertebral level by adding 10-15 mg bupivacaine with 100 μg of morphine.
  Interventions: Drug: Intrathecal bupivacaine and morphine
- Group P+M (Active Comparator): Patients will undergo ultrasound-guided block using a linear or convex ultrasound probe in the supine position before intrathecal bupivacaine plus morphine. The block procedure will involve the use of a local anesthetic solution (10-20 ml of 0.25% bupivacaine and 2 mg dexamethasone) and a 22 Gauche 80 mm block needle. Intrathecal drugs will be administered at the L3-L4 intervertebral level by adding 10-15 mg bupivacaine with 100 μg of morphine.
  Interventions: Drug: Pericapsular nerve group block plus intrathecal bupivacaine and morphine

INTERVENTIONS:
Drug: Pericapsular nerve group block plus intrathecal bupivacaine — Patients will undergo ultrasound-guided block using a linear or convex ultrasound probe in the supine position before intrathecal bupivacaine. The block procedure will involve the use of a local anesthetic solution (10-20 ml of 0.25% bupivacaine and 2 mg dexamethasone) and a 22 Gauche 80 mm block needle. Subsequently, intrathecal bupivacaine will be administered at the L3-L4 intervertebral level with 10-15 mg bupivacaine while the patient is in a sitting position.The patient controlled analgesia device with morphine will be adjusted as infusion: 0 ml/h, bolus: 1 mg/h, lockout period: 10 min.
  Other Names: Spinal anesthesia; Peripheric nerve block
  Arms: Group P
Drug: Intrathecal bupivacaine and morphine — Patients will receive intrathecal bupivacaine and morphine without Pericapsular Nerve Group block. Intrathecal drugs will be administered at the L3-L4 intervertebral level by adding 10-15 mg bupivacaine with 100 μg of morphine. The patient controlled analgesia device with morphine will be adjusted as infusion: 0 ml/h, bolus: 1 mg/h, lockout period: 10 min.
  Other Names: Spinal anesthesia
  Arms: Group M
Drug: Pericapsular nerve group block plus intrathecal bupivacaine and morphine — Patients will undergo ultrasound-guided block using a linear or convex ultrasound probe in the supine position before intrathecal drugs. The block procedure will involve the use of a local anesthetic solution (10-20 ml of 0.25% bupivacaine and 2 mg dexamethasone) and a S22 Gauche 80 mm block needle. Subarachnoid block will be administered at the L3-L4 intervertebral level by adding 10-15 mg bupivacaine with 100 μg of morphine. The patient controlled analgesia device with morphine will be adjusted as infusion: 0 ml/h, bolus: 1 mg/h, lockout period: 10 min.
  Other Names: Spinal anesthesia; Peripheric nerve block
  Arms: Group P+M

SUMMARY:
This study aims to compare the postoperative 48-hour period in terms of morphine consumption, postoperative pain, and quality of recovery scores by combining the Pericapsular Nerve Group (PENG) block with low-dose intrathecal morphine in hip arthroplasty, as opposed to PENG alone and intrathecal morphine alone.

DETAILED DESCRIPTION:
Effective postoperative pain control in hip surgeries can reduce complications and improve postoperative care. Multimodal analgesic techniques in postoperative pain management are employed to synergistically target different nociceptive mechanisms. Combining peripheral nerve blocks with low-dose intrathecal opioids can decrease the systemic opioid dose. Additionally, side effects associated with opioids, such as sedation, respiratory depression, nausea, vomiting, rash, and urinary retention, can be mitigated by the combination with peripheral nerve blocks.

The addition of Pericapsular Nerve Group (PENG) block to a multimodal analgesia regimen has been shown to significantly enhance the quality of recovery and reduce opioid consumption in patients undergoing hip arthroplasty.

The Quality of Recovery (QoR-15), developed and validated by Stark et al. in 2013, is a recovery scale indicating postoperative recovery quality. It includes 15 questions assessing pain, physical comfort, physical independence, psychological support, and emotional state, providing a score between 0 and 150, where a higher score indicates better recovery quality.

In anterior hip surgeries, it is anticipated that spinal anesthesia combined with PENG block and low-dose intrathecal morphine will result in lower postoperative morphine consumption and pain scores compared to PENG alone and intrathecal morphine alone over the first 48 hours. Furthermore, it is expected that the quality of recovery (QoR-15 score) will be higher, providing patients with a longer pain-free period, early mobilization, and improved recovery quality.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 90 years
* American Society of Anesthesiologists (score ranging from 1 to 4)
* Anterior hip arthroplasties

Exclusion Criteria:

* Patients with a history of opioid addiction
* Individuals under the age of 18
* Those aged 90 and above
* Allergies to morphine, fentanyl, bupivacaine, or tramadol
* Coagulopathy
* Infection at the injection site
* Severe cardiac, renal, or hepatic dysfunction
* Cases unable to provide informed consent
* Body Mass Index >40 kg/m2
* Known neurological or anatomical deficits in the lower extremities
* Patients requiring a transition from spinal anesthesia to general anesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-03-18 (Estimated); Primary Completion 2024-06-08 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | From end of anesthesia (15 minutes after anesthesia) to after 48 hours, up to 48 hours
  Morphine

SECONDARY OUTCOMES:
Postoperative pain scores | From end of anesthesia (15 minutes after anesthesia) to after 48 hours, up to 48 hours
  Visual Analog Scale (Minimum value: 0- Maximum value:10) 0: No pain, 10: the most intense pain imaginable. Lower scores mean better outcomes and higher scores mean worse outcome.
The quality of recovery score | From beginning of anesthesia (15 minutes before anesthesia) to after 24 hours, up to 24hours
  The quality of recovery (QoR-15 score): It includes 15 questions assessing pain, physical comfort, physical independence, psychological support, and emotional state, providing a score between 0 and 150, where a higher score indicates better recovery quality.

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Oztop, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT06298370/Prot_SAP_000.pdf